CLINICAL TRIAL: NCT06264817
Title: A Multicenter, Single-blinded, Randomized Controlled Study to Assess the Efficacy of Auto-Adjustable MOBIDERL Autofit Armsleeve in the Management of Upper Limb Lymphedema. (LyberT)
Brief Title: Auto-Adjustable MOBIDERm Autofit Armsleeve in the Management of Upper Limb Lymphedema.
Acronym: LyberT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 48 LyberT
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Lymphedema of Upper Limb
Keywords: Lymphedema of upper limb; Compression garments; lymphedema management

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, interventional, controlled-randomized, single blinded study
Who Masked: Outcomes Assessor
Masking Description: For the same patient, all measurements will be performed as far as possible by the same health professional who doesn't have the knowledge of patient's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group : compressive bandaging (Active Comparator): Control group : compressive bandaging:
  * Intensive phase (3 weeks): compressive bandaging (day and night-time) according to the usual practice
  * Maintenance phase (5 weeks): usual compression sleeve during the day + Self bandages at night
  Interventions: Device: Compressive bandaging
- Intervention group: MOBIDERM Autofit Armsleeve (Experimental): Intervention group: MOBIDERM Autofit Armsleeve
  * Intensive phase (3 weeks): MOBIDERM Autofit Armsleeve (day and night-time)
  * Maintenance phase (5 weeks): usual compression sleeve during the day + MOBIDERM Autofit Armsleeve at night
  Interventions: Device: MOBIDERM Autofit Armsleeve

INTERVENTIONS:
Device: MOBIDERM Autofit Armsleeve — In the intervention group, during the intensive phase, patients wear day and night MOBIDERM AUTOFIT during 3 weeks.
  During the maintenance phase, patients wear usual compression sleeve during the day and MOBIDERM Autofit Armsleeve at night during 5 weeks
  Arms: Intervention group: MOBIDERM Autofit Armsleeve
Device: Compressive bandaging — In the control group, during the intensive phase, patients wear compressive bandaging day and night-time, according to the usual practice during 3 weeks.
  During the maintenance phase, patients wear usual compression sleeve during the day and self bandages at night during 5 weeks
  Arms: Control group : compressive bandaging

SUMMARY:
This study aims to assess Auto-Adjustable MOBIDERM® Autofit Armsleeve effect on upper limb volume excess compared to the compression bandages to manage the volume of upper limb lymphedema in patients with breast cancer related lymphedema

DETAILED DESCRIPTION:
The overall range of compression devices dedicated to lymphedema treatment offers standard or custom-made garments and different types of bandages. Indeed, bandages are not easy to put on, requiring specific patient's skills and/or assistance which is not optimal for long-term compliance. Moreover, they are composed of several layers forming a quite bulky multilayer bandage that limits limb function and does not contribute to a better quality of life. For all these reasons described, even if bandaging is the current reference of lymphedema treatment, they have disadvantages.

The day-time elastic compressive armsleeves are proposed as an alternative to bandages. However, whatever their standard or custom-made design, they cannot adapt to limb volume/morphology evolution on the long-term management of this chronic disease because they are not adjustable. Therefore, as the comfort of treatment is very important in improving compliance, armsleeves are sometimes poorly tolerated by patients resulting in decreasing compliance to treatment plan.

In order to optimize treatment of lymphedema efficacy, THUASNE developed the standard Auto-Adjustable Armsleeve using the MOBIDERM technology.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral secondary upper limb lymphedema of stage II or III according to the criteria defined by the International Society of Lymphology, following breast cancer
* Volume difference between affected and healthy arm ≥ 10%
* Affected arm that fits with one of the 6 standard sizes of the Auto- Adjustable MOBIDERM Autofit armsleeve provided.
* Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

* Stage I lymphedema or located in several places.
* Patients for whom compression is contraindicated.
* Lymphedema associated with active cancer needing acute chemotherapy or having recurrence or metastasis.
* Motor and sensitive neurological deficiency / psychiatric or addictive disorders
* Pregnant or breastfeeding patient
* Patient intolerant to MOBIDERM Autofit or known allergies to the components used.
* Participation to any other clinical study which has an impact on the different endpoints
* Vulnerable patient, adults being the object of a legal protective measure or enable to express their consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Volume excess variation | 8 weeks
  The primary endpoint of this study is to compare between both groups the volume evolution of the upper limb between inclusion and the end of the study. Limb Volume is calculated with truncated cone formula.

SECONDARY OUTCOMES:
Resource consumption | 3 and 8 weeks
  Resource consumption is measured by time of transports (travel time in minutes).
Resource consumption | 3 and 8 weeks
  Resource consumption is measured by number of used medical devices (number).
Resource consumption | 3 and 8 weeks
  Resource consumption is measured by the number and duration (per minute) of lymphedema-related healthcare consultations and hospitalizations.
Lymphedema related Quality of life (QoL) | 3 and 8 weeks
  The evolution of QoL is measured by LYMQOL ARM self-questionnaire and specific questions. This tool is designed as patient-completed questionnaire. The questions cover four domains : symptoms, body image/appearance, function, mood. Each item in each domain is scored : not at all (1), a little (2), Quite a bit (3), A lot (4). Specific questions are about patient's perception of benefit
Doctors' opinion on improving the patient's health condition | 3 and 8 weeks
  Doctors' opinion on improving the patient's health condition caused by lymphedema is measured by the CGI-I questionnaire (Clinical Global Improvement Impression). This questionnaire allows doctors to evaluate the improvement of patients. The scale has 7 levels from "very strongly improved"(better outcome) to "very strongly aggravated"(worse outcome).Intermediate levels are: " Significantly improved " ; " Slightly improved " ; " No improvement " ; " Slightly aggravated " ; " Seriously aggravated "
Patient's opinion on Global Impression of Change | 3 and 8 weeks
  Patient's opinion on Global Impression of Change about her general condition is measured by the PGI-C questionnaire (Patient's opinion on Global Impression of Change). The scale has 7 levels from "no change or condition has got worsed"(worse outcome) to "a great deal better, and a considerable improvement that has made all the difference ( better outcome)". Intermediate levels are: "almost the same, hardly any change at all"; "a little better, but no noticeable change", "somewhat better, but the change has not made any real difference"; "moderately better, and a slight but noticeable change"; "better, and a definite improvement that has made a real and worthwhile difference
Satisfaction about the device | 8 weeks
  Patient's satisfaction with regards to MOBIDERM® Autofit vs bandages is measured by a satisfaction questionnaire. This questionnaire is focused on the product positioning with a question with 4 levels: very easy (better outcome), easy, difficult, very difficult (worse outcome) and the comfort with a question with 4 levels very comfortable (better outcome), comfortable, uncomfortable, very uncomfortable (worse outcome).
The safety | 8 weeks
  Number and type of serious and non-serious Adverse Device Effects (ADE).
Compliance to treatment | 8 weeks
  The compliance to treatment (day-time and night-time) is reported by the physician in the e-CRF according to the patient diary. The compliance is measured in number of days and or nights when the device is worn and the average wearing time
General quality of life (QoL) | 3 and 8 weeks
  The evolution of QoL is measured by the EQ5D3L questionnaire completed by the patient. The EQ-5D3L questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems (Level 1 is coded as a '1'), moderate problems (Level 2 is coded as a '2'), and extreme problems (Level 3 is coded as a '3'). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS). The EQ VAS is measured by VAS : 100 corresponds to the best health and 0 to the the worst health.
Skin elasticity | 3 and 8 weeks
  The evolution of skin thickness and elasticity is measured by ultrasound
Ttissue induration | 3 and 8 weeks
  The evolution of tissue induration is measured via the skinfibrometer (Delfin Tech).

CONTACTS AND LOCATIONS:
Overall Officials: Burcu DUYUR ÇAKIT, Principal Investigator — Ankara Training and Research Hospital Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - ANKARA, Ankara
  - Pinar BORMAN, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ochalek K, Kurpiewska J, Gradalski T. Adjustable Compression Wraps (ACW) vs. Compression Bandaging (CB) in the Acute Phase of Breast Cancer-Related Arm Lymphedema Management-A Prospective Randomized Study. Biology (Basel). 2023 Mar 31;12(4):534. doi: 10.3390/biology12040534. PMID 37106735
- [Background] Mestre S, Calais C, Gaillard G, Nou M, Pasqualini M, Ben Amor C, Quere I. Interest of an auto-adjustable nighttime compression sleeve (MOBIDERM(R) Autofit) in maintenance phase of upper limb lymphedema: the MARILYN pilot RCT. Support Care Cancer. 2017 Aug;25(8):2455-2462. doi: 10.1007/s00520-017-3652-5. Epub 2017 Mar 9. PMID 28281052
- [Background] Borman P, Koyuncu EG, Yaman A, Calp E, Koc F, Sargut R, Karahan S. The Comparative Efficacy of Conventional Short-Stretch Multilayer Bandages and Velcro Adjustable Compression Wraps in Active Treatment Phase of Patients with Lower Limb Lymphedema. Lymphat Res Biol. 2021 Jun;19(3):286-294. doi: 10.1089/lrb.2020.0088. Epub 2020 Dec 2. PMID 33270499